CLINICAL TRIAL: NCT03378037
Title: The Effects of Acupuncture on the Risk of AD After TBI: A Randomized Controlled Trial
Brief Title: The Effects of Acupuncture on the Risk of AD After TBI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUH106-REC2-139
Record Dates: First submitted 2017-12-08; First posted 2017-12-19 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Brain Injuries, Traumatic
Keywords: Brain Injuries, Traumatic; Alzheimer's disease; Magnetic resonance imaging; white matter integrity; beta-Amyloid
MeSH Terms: conditions — Brain Injuries, Traumatic; Alzheimer Disease; Plaque, Amyloid | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture group (Experimental): Disposable acupuncture needles will be inserted into acupoints for a depth of 10-30 mm in a direction oblique or parallel to the surface. To ensure allocation concealment, all needles will be affixed with plastic O-rings and adhesive tapes.
  Interventions: Procedure: Acupuncture
- Control group (Sham Comparator): Streitberger's non-invasive placebo acupuncture needles will be used in the control group; blunt-tipped needles will touch the skin quickly without being inserted. To ensure allocation concealment, all needles will be affixed with plastic O-rings and adhesive tapes.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — 20 minutes of acupuncture treatment, twice a week for 2 weeks. Acupoints will be manually stimulated every 10 minutes.

SUMMARY:
Traumatic brain injury (TBI) is a severely disabling injury which affects 150-200 people per million annually. Increasing evidence suggests that TBI may be a major risk of dementia, Alzheimer's disease (AD) in particular. Postmortem evidence has shown that beta-amyloid (Aβ) deposits, one of the most validated pathological biomarkers of AD, are present in the brains of severe TBI patients. Although the underlying mechanisms remain unclear, the axonal injury may play a role. Imaging investigations have revealed Aβ density maps of TBI patients overlapped with those of AD patients, and increased Aβdensity not only associated with prolonged TBI duration but also associated with decreased white matter integrity. Hence, the increasing accumulation in Aβ due to TBI may contribute to the initiation of the pathological alterations seen in AD. Treatment of TBI may not only be of benefit for the injury itself but also act to block the pathological changes in AD.

As a part of the clinical arm of the project, in this subproject investigators will conduct a single-blind, block-randomized clinical trial to investigate the efficacy of acupuncture in TBI. More specifically, investigators hypothesize that acupuncture intervention will elicit neuroprotective processes and thereby reduce axonal damage in TBI, manifested as (1) decreased plasma levels of Aβ peptide, tau, and glial fibrillary acidic protein (GFAP) and (2) increased white matter integrity after acupuncture. Ninety-six participants will be randomly allocated to the acupuncture intervention (verum acupuncture) or control group (sham acupuncture) in a 1:1 ratio. All participants will receive 20 minutes of acupuncture treatment twice a week for 2 weeks. A set of commonly used acupoints for TBI treatment will be manually stimulated every 10 minutes. The multi-modality magnetic resonance imaging (T1, T2, and diffusion tensor imaging) and blood sample will be taken before and after the acupuncture session to measure the white matter integrity in brain and plasma levels of Aβ peptide, tau, and GFAP, respectively. After integrate these data with other subprojects, we can provide synergic and integrative mechanisms of the effects of acupuncture on the risk of AD after TBI.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 20 years old
2. GCS score > 13
3. LOC < 30 minutes
4. hospital admission < 7 days
5. having adequate competency for understanding the study and a willingness to sign the written informed consent forms
6. be able to commence the acupuncture intervention within 2 weeks after TBI diagnosis

Exclusion Criteria:

1. medical history of neurological, cardiovascular events, or mental disorder, e.g., epilepsy, stroke, major depression or anxiety
2. other major medical conditions, e.g., active cancer, uncontrolled diabetes, pregnancy
3. surgery for TBI
4. receipt of acupuncture within the 6 months prior to study entry
5. patients with pacemaker, metal graft, or claustrophobia
6. preparing for pregnancy during the trial

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2017-12-25 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Decreased plasma levels of Aβ peptide | After 2-week acupuncture treatment interval
Decreased plasma levels of tau | After 2-week acupuncture treatment interval
Decreased plasma levels of glial fibrillary acidic protein (GFAP) | After 2-week acupuncture treatment interval

SECONDARY OUTCOMES:
Increased white matter integrity | After 2-week acupuncture treatment interval

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan